CLINICAL TRIAL: NCT04098458
Title: Single-Arm Trial Assessing the Feasibility and Acceptability of Navigation for The Management of Delays and Racial Disparities Starting Adjuvant Therapy in Adults With Surgically-Managed, Locally Advanced HNSCC (NDURE 2.0 Pilot)
Brief Title: Navigation for Timely Adjuvant Therapy for Patients With Locally Advanced HNSCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Graboyes, Assistant Professor, Department of Otolaryngology-Head & Neck Surgery, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00091049-A; K08CA237858 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NDURE (Experimental): NDURE is a navigation-based, multilevel intervention targeting barriers to timely, guideline-adherent PORT at the patient-, healthcare team-, and organization-levels.
  Interventions: Behavioral: NDURE

INTERVENTIONS:
Behavioral: NDURE — NDURE consists of 6 key functions including (1) Improve patient knowledge about guidelines for timely PORT and associated care processes; (2) Minimize the burden of travel for HNSCC care; (3) Improve communication between patients and providers regarding intentions and goals for timely, guideline-adherent PORT; (4) Enhance coordination of care between healthcare teams during care transitions and about treatment sequelae; (5) Track referrals to ensure timely scheduling of appointments and patient attendance across fragmented healthcare systems; (6) Restructure the organization to clarify roles and responsibilities for care processes associated with PORT delivery to avoid duplication and gaps in care. Direct contact between the NDURE navigator and patient occurs via three clinic-based, face-to-face NDURE sessions lasting 30-60 minutes each at the pre-surgical consult, hospital discharge, and first postoperative visit.

SUMMARY:
Head and neck cancer squamous cell carcinoma (HNSCC) is a disease with poor survival, especially for African Americans, despite intense treatment including surgery, radiation, and chemotherapy. Delays between surgery and the start of postoperative radiation therapy (PORT) are common, cause excess mortality, and contribute to worse survival in African Americans. Our research team has developed NDURE (Navigation for Disparities and Untimely Radiation thErapy), a novel theory-based patient navigation (PN) intervention to decrease delays and racial disparities starting PORT. In this single-site, open label, single-arm trial, adults with surgically-managed, locally advanced HNSCC, will be enrolled in NDURE to assess the feasibility and acceptability of NDURE as a novel approach to decreasing delays and racial disparities starting PORT after surgery for HNSCC. The investigators will collect information about the accrual rate and NDURE completion rate. Participants will also complete validated questionnaires at baseline and post-intervention to evaluate the feasibility of outcome assessment for NDURE. Post-intervention, patients and providers will undergo interviews to obtain in-depth understanding of the content, format, timing, and delivery of NDURE to optimize the intervention in preparation for a future multi-site study. NDURE could provide the first effective intervention to improve the delivery of timely, equitable PORT after HNSCC surgery, thereby improving survival for patients with HNSCC, decreasing racial disparities in mortality, and developing new standards of clinical care.

DETAILED DESCRIPTION:
Design: The study design is a single-site, single-arm, trial of NDURE (Navigation for Disparities and Untimely Radiation thErapy) to assess the feasibility and acceptability of this patient navigation (PN) intervention to decrease delays and racial disparities starting postoperative radiation therapy (PORT) after surgery for HNSCC.

Following screening and informed consent, sociodemographic and oncologic will be prospectively gathered about participants from validated questionnaires and the electronic medical record (EMR). Participants will undergo 3 sessions of NDURE. Measures of feasibility (enrollment, dropout, missed PN encounters, navigator caseload, and time allocation) will be assessed during delivery of NDURE. Questionnaires assessing symptom burden and health-related beliefs will be collected at baseline and post-treatment to assess the feasibility of data collection procedures and monitor completion rates. Following completion of NDURE, patients with HNSCC will complete validated measures of acceptability related to satisfaction with PN. Post-NDURE qualitative work with patients and providers will help refine the intervention

Treatment Allocation: Participants will be enrolled into NDURE

Delivery of intervention: NDURE is a navigation-based, multilevel intervention targeting barriers to timely, guideline-adherent PORT at the patient-, healthcare team-, and organization-levels. NDURE consists of 6 key functions including (1) Improve patient knowledge about Guidelines for timely PORT and associated care processes; (2) Minimize the burden of travel for HNSCC care; (3) Improve communication between patients and providers regarding intentions and goals for timely, guideline-adherent PORT; (4) Enhance coordination of care between healthcare teams during care transitions and about treatment sequelae; (5) Track referrals to ensure timely scheduling of appointments and patient attendance across fragmented healthcare systems; (6) Restructure the organization to clarify roles and responsibilities for care processes associated with PORT delivery to avoid duplication and gaps in care.

Direct contact between the NDURE navigator and patient occurs via three clinic-based, face-to-face NDURE sessions lasting 30-60 minutes each. The three NDURE sessions coincide with the pre-surgical consult, hospital discharge, and first postoperative visit, time points chosen to facilitate case identification and coordination across care transitions. During each NDURE session, the navigator delivers patient education and creates or updates the PORT Care Plan. Referral tracking and follow-up occurs through asynchronous contact between the navigator, patient, and healthcare organizations between NDURE sessions.

The sample size justification for this single-arm study is based on the primary feasibility endpoints of NDURE accrual and completion. In the randomized controlled trial (RCT) of NDURE (NCT04030130), the investigators plan to enroll 60% of eligible patients. The investigators expect similar accrual in this feasibility study and therefore, accruing to NDURE will be considered feasible if at least 15 of 25 eligible subjects enroll. Our sample size was selected to provide a small probability of having an observed accrual rate of at least 60% when the true accrual probability is actually less than 60%. For example, if the true accrual probability for our proposed design is 45% (35%), the probability of enrolling 15 or more of 25 eligible subjects is only 10% (1%). Additionally, the investigators target an NDURE completion rate ≥85%. That is to say, NDURE is feasible if at least 13 of the 15 subjects enrolled complete all three in-person NDURE sessions. Accordingly, the sample size for the single-arm study was selected to provide a small probability of having an observed completion rate of at least 85% when the true completion probability of the intervention is actually less than 85%. For example, if the true completion probability for our proposed design is 70% (60%), the probability that 13 or more of the 15 enrolled patients complete all three in-person NDURE sessions is 13% (3%). Therefore, the probability of falsely declaring NDURE feasible is reasonably controlled based on this sample size.

Statistical Methods of Analysis: This aim is descriptive, and the statistical analysis focuses on characterizing the feasibility and acceptability of NDURE. To examine patterns and characterize sociodemographic, oncologic, and symptom burden variables, the investigators will construct graphical displays and descriptive statistics (e.g. frequencies and percent for categorical variables and mean, median, standard deviation, and range for continuous variables). Feasibility measures for study accrual rate will evaluate the proportion and frequency of eligible patients who accrue (overall, white, and African American). Given its pilot nature, the study is not designed to evaluate racial differences in accrual, although reasons for study decline will be collected, analyzed for each racial subgroup, and used to refine recruitment. NDURE completion rate will be analyzed as 1) the percentage of enrolled patients who attend all three in-person NDURE sessions and 2) the proportion of three in-person NDURE sessions that are completed. For navigator caseload, the investigators will consider the frequency of simultaneous cases navigated. Navigator time allocation for direct and indirect time, as well as patient-report measures of satisfaction with navigation will be summarized as described above for continuous data. Study questionnaire completion rate will be calculated as the proportion of pre- and post-intervention questionnaires (n=5 each) completed. Qualitative data will be analyzed using established team codebooks and focus on the content, format, delivery, and timing of NDURE. Qualitative analysis of semi-structured interviews with patients and providers following the pilot will be analyzed using established codebooks from the study team for evaluating the feasibility and acceptability of clinic-based interventions with a focus on the content, format, delivery, and timing of NDURE.

ELIGIBILITY:
Inclusion Criteria:

Patient and disease characteristics

1. Age > 18 years at the time of screening
2. Histologically or pathologically confirmed invasive SCC (or histologic variant) of the oral cavity, oropharynx (p16 positive, negative, or unknown), hypopharynx, larynx, unknown primary, paranasal sinuses, or nasal cavity.

   a. In situations in which the patient fulfills all other inclusion criteria but the biopsy shows SCC in-situ or moderate/severe dysplasia (without definitive evidence of invasive SCC), but the patient is scheduled to undergo curative intent surgery by the treating oncologic surgeon due to clinical suspicion of invasive SCC, the diagnosis of SCC-in situ or moderate/severe dysplasia is sufficient to full the pathologic diagnosis enrollment criterion.
3. American Joint Committee on Cancer (AJCC) clinical stage grouping III-IV (8th edition) for patients with SCC of the oral cavity, p16-negative oropharynx, hypopharynx, larynx, paranasal sinuses, and nasal cavity; or AJCC clinical stage grouping III-IV (7th edition) for patients with p16-positive SCC of the oropharynx or unknown primary.

   1. At screening, AJCC clinical stage grouping should be determined based on a combination of physical exam, diagnostic evaluation with cross sectional imaging of the neck (computerized tomography (CT) and/or magnetic resonance imaging (MRI)) and/or 18-F-fluoro-deoxyglucose positron emission tomography (FDG PET) CT within 30 days
   2. In situations in which the patient fulfills all other inclusion criteria but the biopsy shows SCC in-situ or moderate/severe dysplasia (without definitive evidence of invasive SCC), but would otherwise have an appropriate clinical stage grouping as defined in criterion 5, the diagnosis of SCC-in situ or moderate/severe dysplasia is sufficient to full the staging enrollment criterion.
4. No prior exposure to radiation therapy, with or without concurrent chemotherapy, for treatment of HNSCC in the definitive or adjuvant therapy settings

   Surgery and adjuvant therapy eligibility
5. Plan for curative intent surgery at MUSC

   a. At screening, plan for curative intent surgical resection of the HNSCC at MUSC must be deemed likely by the treating surgeon and/or multidisciplinary tumor board, which must include a fellowship-trained head and neck oncologic surgeon
6. Plan for PORT (at MUSC or non-MUSC) with or without concurrent chemotherapy following curative intent surgery a. At screening, plan for adjuvant therapy following curative intent surgical resection of the HNSCC at MUSC must be deemed likely by the treating surgeon and/or multidisciplinary tumor board, which must include a fellowship-trained head and neck oncologic surgeon, based on the clinical expectation of at least one of the following adverse features on final pathologic evaluation: extranodal extension (ENE), pathologic T3 or T4 primary, N2 or N3 nodal disease, nodal disease in levels IV or V, perineural invasion (PNI), or lymphovascular invasion (LVI)

Exclusion Criteria:

1. Self-identified Hispanic ethnicity
2. Presence of cognitive impairment that precludes participation
3. Failure to undergo curative intent surgery at MUSC
4. Lack of indication for PORT (with or without concurrent chemotherapy) per National Comprehensive Cancer Network (NCCN) Guidelines based on the presence of at least one of the following adverse features on final pathologic evaluation: ENE, positive margin, pathologic stage T3 or T4 primary, pathologic stage N2 or N3 nodal disease, nodal disease in levels IV or V, perineurial invasion, or lymphovascular invasion
5. Synchronous untreated malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NDURE: Navigation for Disparities and Untimely Radiation thErapy (NDURE) is a navigation-based, multilevel intervention targeting barriers to timely, guideline-adherent postoperative radiation therapy (PORT). NDURE key functions include: 1) Improve patient knowledge about Guidelines for timely PORT and associated care processes; 2) Minimize the burden of travel for HNSCC care; 3) Improve communication between patient and providers regarding intentions and goals for timely, guideline-adherent PORT; 4) Enhance care coordination between care teams during care transitions and about treatment sequelae; 5) Track referrals to ensure timely scheduling of appointments and patient attendance across fragmented healthcare systems; 6) Restructure the organization to clarify roles and responsibilities for care processes associated with PORT delivery to avoid duplication and gaps in care.
  Direct contact between the NDURE navigator and patient occurs via three clinic-based, face-to-face NDURE sessions lasting 30-60 minutes each. The three NDURE sessions coincide with the pre-surgical consult, hospital discharge, and first postoperative visit, time points chosen to facilitate case identification and coordination across care transitions. During each NDURE session, the navigator delivers patient education and creates or updates the PORT Care Plan. Referral tracking and follow-up occurs through asynchronous contact between the navigator, patient, and healthcare organizations between NDURE sessions.
Period: Overall Study
Arm/Group | NDURE
Started | 18
Completed | 14
Not Completed | 4
Not completed — Death | 1
Not completed — did not meet study inclusion criteria | 3

BASELINE CHARACTERISTICS:
Arm/Group | NDURE
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Health Insurance Coverage [Count of Participants; unit: Participants]
  Private | 6
  Medicare | 6
  Medicaid | 1
  Self-pay | 2
Marital Status [Count of Participants; unit: Participants]
  Married/current partner | 8
  Single/separated/divorced/widowed | 7
Living Situation [Count of Participants; unit: Participants]
  Spouse/partner | 7
  Parents/siblings/children | 3
  Self | 5
Highest Level of Education [Count of Participants; unit: Participants]
  High school graduate | 5
  Some college | 4
  College or graduate school | 6
Employment [Count of Participants; unit: Participants]
  Full or part-time paid | 5
  Retired | 7
  Disability or unemployed | 3
Subsite [Count of Participants; unit: Participants]
  oral cavity | 13
  Oropharynx (human papillomavirus-related) | 1
  Paranasal sinus | 1
American Joint Committee on Cancer Pathologic T Category [Count of Participants; unit: Participants] — Patients were staged using the American Joint Committee on Cancer (AJCC) 8th Edition Staging Manual for Head and Neck Cancer. Pathologic T category is determined by pathologic evaluation of the main cancer specimen following surgery. Pathologic T category ranges from 0 to 4b, with higher AJCC T category representing more locally advanced head and neck cancer
  Participants
    1-2 | 2
    3-4b | 13
American Joint Committee on Cancer Pathologic N Category [Count of Participants; unit: Participants] — Patients were staged using the American Joint Committee on Cancer (AJCC) 8th Edition Staging Manual for Head and Neck Cancer. Pathologic N category is determined by pathologic evaluation of the lymph nodes from the neck dissection specimen following surgery. Pathologic N category ranges from 0 to 3b, with higher AJCC N category representing more regionally advanced head and neck cancer
  Participants
    0-1 | 11
    2-3b | 4
Overall American Joint Committee on Cancer Stage Grouping [Count of Participants; unit: Participants] — Patients were staged using the American Joint Committee on Cancer (AJCC) 8th Edition Staging Manual for Head and Neck Cancer. Overall AJCC Pathologic Stage Grouping is determined by combining the pathologic T, N, and M categories. Overall pathologic AJCC Stage Grouping ranges from 0 to IVc, with higher stage grouping representing more advanced head and neck cancer
  Participants
    III | 1
    IV | 14
Adjuvant Therapy [Count of Participants; unit: Participants] — Population: 1 participant suffered a mortality prior to initiating adjuvant radiation and the measure is thus not analyzable for this participant
  Participants
    number analyzed (Participants) | 14
    Radiation | 7
    Chemoradiation | 6
    Immuno-radiation | 1
Fragmentation of Care Between Surgical and Radiation Facilities [Count of Participants; unit: Participants] — Population: 1 participant suffered a mortality prior to initiating adjuvant radiation and the measure is thus not analyzable for this participant
  Participants
    number analyzed (Participants) | 14
    No | 7
    Yes | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Participants Who Accrue to NDURE
Description: Percent of eligible participants who accrue to NDURE, defined as a participant who meets all inclusion criteria and no exclusion criteria
Time Frame: 5 months
Population: percentage of participants meeting all inclusion/exclusion criteria who accrued to the study
Measure: Count of Participants; unit: Participants
Arm/Group | NDURE
Number analyzed (Participants) | 17
Participants | 15

2. Secondary Outcome: Percent of Participants Who Complete the NDURE Intervention and Study Measures
Description: Completion of the baseline assessment, at least two (of 3) NDURE intervention sessions, and the end of study assessment
Time Frame: 5 months
Population: intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- NDURE: NDURE is a navigation-based, multilevel intervention targeting barriers to timely, guideline-adherent PORT at the patient-, healthcare team-, and organization-levels. NDURE consists of 6 key functions including (1) Improve patient knowledge about Guidelines for timely PORT and associated care processes: (2) Minimize the burden of travel for HNSCC care; (3) Improve communication between patient and providers regarding intentions and goals for timely, guideline-adherent PORT; (4) Enhance coordination of care between healthcare teams during care transitions and about treatment sequelae; (5) Track referrals to ensure timely scheduling of appointments and patient attendance across fragmented healthcare systems; (6) Restructure the organization to clarify roles and responsibilities for care processes associated with PORT delivery to avoid duplication and gaps in care.
  Direct contact between the NDURE navigator and patient occurs via three clinic-based, face-to-face NDURE sessions lasting 30-60 minutes each. The three NDURE sessions coincide with the pre-surgical consult, hospital discharge, and first postoperative visit, time points chosen to facilitate case identification and coordination across care transitions. During each NDURE session, the navigator delivers patient education and creates or updates the PORT Care Plan. Referral tracking and follow-up occurs through asynchronous contact between the navigator, patient, and healthcare organizations between NDURE sessions.
Arm/Group | NDURE
Number analyzed (Participants) | 15
Participants | 14

3. Secondary Outcome: Satisfaction With the Interpersonal Relationship With the Navigator (PSN-I) Scale Score
Description: The PSN-I measures the satisfaction with the interpersonal relationship with the patient navigator. The PSN-I score is defined as the total score of this 9-item scale. The total score ranges from 9 (minimum) to 45 (maximum); higher scores represent a better outcome (greater satisfaction with the interpersonal relationship with the navigator).
Time Frame: Post-intervention (3 months)
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 38 (2.9)

4. Secondary Outcome: Navigator Caseload
Description: The number of simultaneous cases (on-trial participants) being navigated by the NDURE navigator
Time Frame: 5 months
Population: ITT
Measure: Mean (Full Range); unit: simultaneous cases
Arm/Group | NDURE
Number analyzed (Participants) | 15
simultaneous cases | 3.5 [1 to 5]

5. Secondary Outcome: Navigator Time Allocation (Direct)
Description: The time (in minutes), that the NDURE navigator spends directly interacting with the patient to identify and address barriers to timely, equitable postoperative radiation therapy.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Full Range); unit: minutes per patient
Arm/Group | NDURE
Number analyzed (Participants) | 14
minutes per patient | 96 [90 to 135]

6. Secondary Outcome: Navigator Time Allocation (Indirect)
Description: The time (in minutes), that the navigator spends generating and enacting each Barrier Reduction Plan that is not directly interacting with the patient
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure.
Measure: Mean (Full Range); unit: minutes/patient
Arm/Group | NDURE
Number analyzed (Participants) | 14
minutes/patient | 135 [120 to 195]

7. Secondary Outcome: Navigator Time Allocation (Total)
Description: The time (in minutes), that the NDURE navigator spends directly or indirectly interacting with the patient to identify and address barriers to timely, equitable postoperative radiation therapy
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Full Range); unit: minutes/patient
Arm/Group | NDURE
Number analyzed (Participants) | 14
minutes/patient | 231 [210 to 330]

8. Secondary Outcome: Percent of Patients With a Delay Starting Post-Operative Radiation Treatment
Description: Percent of patients who start PORT >6 weeks after surgery. Initiation of postoperative PORT > 6 weeks after surgery is defined as more than 42 calendar days from the time of the definitive surgical resection to the initiation of radiation therapy. In situations in which the surgical management of the primary tumor and the neck are staged (i.e. occur on two different calendar days), the date of the surgery for the primary tumor will be used. In situations in which an additional surgical resection is required (e.g. re-resection of positive margins to clear residual disease), the date of the earlier (i.e. attempted definitive) surgical procedure will be used to determine the target start date for PORT.
Time Frame: 6 weeks
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | NDURE
Number analyzed (Participants) | 14
Participants | 2

9. Secondary Outcome: Percent Difference in PORT Delay Between White and Black Patients With Head and Neck Cancer
Description: The difference in the rate of initiation of PORT > 6 weeks after surgery between white and black patients with head and neck cancer (i.e., percent difference = percent of white patients with PORT delay minus percent of black patients with PORT delay)
Time Frame: 6 weeks
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Number; unit: percentage of participants
Arm/Group | NDURE
Number analyzed (Participants) | 14
percentage of participants | 14.2

10. Secondary Outcome: NDURE Program Evaluation Scale Score: Utility of Sessions With the Navigator
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The sessions meeting with the navigator were useful to help prevent a delay starting radiation therapy after surgery." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.79 (0.58)

11. Secondary Outcome: NDURE Program Evaluation Scale Score: Timeline of Activities
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The timeline of activities for starting radiation after surgery was useful." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.85 (0.38)

12. Secondary Outcome: NDURE Program Evaluation Scale Score: Helpful in Identifying Challenges Starting Radiation Therapy
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The navigator was helpful in identifying my specific challenges starting radiation therapy after surgery." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
units on a scale | 4.79 (0.58)

13. Secondary Outcome: NDURE Program Evaluation Scale Score: Helpful in Coming up With a Plan to Solve Challenges Starting Radiation
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The navigator was helpful in coming up with a plan to solve my specific challenges starting radiation therapy after surgery." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.85 (0.38)

14. Secondary Outcome: NDURE Program Evaluation Scale Score: Helpful in Solving Challenges Starting Radiation
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The navigator was helpful in solving my specific challenges starting radiation therapy after surgery." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.69 (0.48)

15. Secondary Outcome: NDURE Program Evaluation Scale Score: Material From Navigator Was Relevant
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "he material that I received from the navigator was relevant in helping me address my challenges starting radiation therapy after surgery." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.64 (0.63)

16. Secondary Outcome: NDURE Program Evaluation Scale Score: Timing of Program
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The timing of the program starting at my surgical consultation (before surgery) worked well for me." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.85 (0.38)

17. Secondary Outcome: NDURE Program Evaluation Scale Score: Method of Delivery
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The method of meeting with the navigator to ensure timely head and neck cancer care (face to face) worked well for me." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 5.0 (0.0)

18. Secondary Outcome: NDURE Program Evaluation Scale Score: Number of Sessions
Description: The study-specific program evaluation scale asks participants to rate their agreement with the following statement on a scale of 1-5: "The number of sessions with the navigator (at least 3) worked well for me." Higher scores represent higher levels of agreement.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.43 (1.09)

19. Secondary Outcome: NDURE Program Evaluation Scale Score: Overall Satisfaction
Description: The study-specific program evaluation scale asks participants to rate their satisfaction with the NDURE program on a scale of 1-5; higher scores represent higher levels of satisfaction.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.92 (0.28)

20. Secondary Outcome: NDURE Program Evaluation Scale Score: Likelihood to Recommend
Description: The study-specific program evaluation scale asks participants to rate their likelihood to recommend this program to someone else with head and neck cancer on a scale of 1-5; higher scores represent a greater likelihood of recommending NDURE.
Time Frame: 3 months
Population: ITT; 1 participant who suffered a mortality prior to the end of the study was not evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NDURE
Number analyzed (Participants) | 14
score on a scale | 4.79 (0.58)

ADVERSE EVENTS:
Time Frame: From accrual in the study (at the initial surgical consultation) to the end of the study of the study for each participant (at the start of adjuvant radiation therapy). This time period is variable for participants but on average is approximately 3 months
Description: This trial is considered to carry a low risk to subjects (i.e. has a "no more than minimal risk" designation). As such, this protocol defines an adverse event (AE) as any undesirable sign, symptom, medical, psychological, social, or emotional reaction that is definitely, probably, or possibly related to the study intervention.
Arm/Group | NDURE
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT04098458/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT04098458/Prot_SAP_001.pdf